CLINICAL TRIAL: NCT04602390
Title: A Phase 1 Study of the Safety and Tolerability of Single and Multiple Doses of ANK-700 in Patients With Relapsing Remitting Multiple Sclerosis
Brief Title: Assessment of ANK-700 in Patients With Relapsing Remitting Multiple Sclerosis
Acronym: MoveS-it
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anokion SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ANK-700-01
Record Dates: First submitted 2020-10-05; First posted 2020-10-26 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis (MS); Relapsing Remitting Multiple Sclerosis
Keywords: Autoimmune; Multiple Sclerosis (MS); Relapsing Remitting MS
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- ANK-700 SAD Cohort 1, 0.3 mg/kg ANK-700 (Experimental): All enrolled patients will receive one dose of 0.3 mg/kg ANK-700
  Interventions: Drug: ANK-700
- ANK-700 SAD Cohort 2, 1.0 mg/kg ANK-700 (Experimental): All enrolled patients will receive one dose of 1.0 mg/kg ANK-700
  Interventions: Drug: ANK-700
- ANK-700 SAD Cohort 3, 3.0 mg/kg ANK-700 (Experimental): All enrolled patients will receive one dose of 3.0 mg/kg ANK-700
  Interventions: Drug: ANK-700
- MAD Cohort 4 0.3 mg/kg ANK-700 or Placebo (Experimental): All enrolled patients will receive three doses of 0.3 mg/kg ANK-700 or placebo
  Interventions: Drug: ANK-700; Drug: Placebo
- MAD Cohort 5 1.0 mg/kg ANK-700 or placebo (Experimental): All enrolled patients will receive three doses of 1.0 mg/kg ANK-700 or placebo
  Interventions: Drug: ANK-700; Drug: Placebo

INTERVENTIONS:
Drug: ANK-700 — Intravenous (IV) infusion
Drug: Placebo — Intravenous (IV) infusion
  Arms: MAD Cohort 4 0.3 mg/kg ANK-700 or Placebo; MAD Cohort 5 1.0 mg/kg ANK-700 or placebo

SUMMARY:
A safety study of ANK-700 in patients with relapsing remitting multiple sclerosis. The study has two parts:

Part A - first in human study in which patients receive a single dose of ANK-700 Part B - patients will receive three doses of either ANK-700 or placebo

DETAILED DESCRIPTION:
Study ANK-700-01 is a Phase 1, FIH study designed to evaluate the safety and tolerability of ANK-700 in patients with relapsing remitting multiple sclerosis (rrms).

An overview of the two parts and proposed dose groups is given below:

Part A (SAD): Patients will receive a single dose of ANK-700. Part B (MAD): Patients will receive three doses of either ANK-700 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RRMS per revised McDonald criteria (2017) with an EDSS score ≤ 6.5 at screening
* Neurologically stable with no evidence of relapse within the 28 days before signing the informed consent form (ICF)
* Either not currently receiving disease modifying MS therapy, or currently using fumarate drugs (dimethyl fumarate or diroximel fumarate)
* Patients must use a highly effective method of birth control or are sterile or postmenopausal as confirmed by study Investigator
* Patient has signed and understands the ICF

Exclusion Criteria:

* Diagnosis of primary progressive MS or secondary progressive MS
* Uncontrolled or significant medical conditions (including active infection or chronic hepatitis) which, in the opinion of the Investigator, preclude participation
* Patients treated with glatiramer acetate, parenteral steroids or adrenocorticotropic hormone, β-interferon, plasma exchange within the 3 months prior to first dose
* Patients treated with sphingosine-1-phospate receptor modulators such as fingolimod, ozanimod, or siponimod within 6 months prior to first dose
* Patients treated with cytotoxic agents (including, but not limited to, cladribine, mitoxantrone, cyclophosphamide, azathioprine, and methotrexate), laquinimod, teriflunomide, or IV gamma globulin within 12 months prior to first dose
* Patients treated with monoclonal antibody therapy (including natalizumab, daclizumab, rituximab, ofatumumab, and ocrelizumab) within 24 months prior to first dose
* Patients previously treated with alemtuzumab, total lymphoid irradiation, mesenchymal stem cell or hematopoietic stem cell transplantation, or tolerance-inducing therapies for MS
* Contraindication to or inability to undergo gadolinium-enhanced magnetic resonance imaging (MRI) scan
* Use of any investigational drug or experimental procedure within previous 6 months that would interfere with the assessment of ANK-700
* Patients who are pregnant or breastfeeding
* Patients receiving any vaccination within 28 days prior to first dose
* Patient does not agree to limit alcohol intake to 2 drink equivalents or less per day during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - North Central Neurology, Cullman, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - UC Health Neurosciences Center, Aurora, Colorado
  - Aqualane Clinical Research, Naples, Florida
  - University of South Florida - Neurology, Tampa, Florida
  - University of Kansas Lander Center on Aging/ Neurology, Kansas City, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Cleveland Clinic, Cleveland, Ohio
  - Jefferson University Hospitals, Philadelphia, Pennsylvania
  - Midlands Neurology & Pain Associates PA, Columbia, South Carolina
  - Advanced Neurosciences Institute, Franklin, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas Health Science Center, Houston, Texas
  - MS Center of Greater Washington, Vienna, Virginia
  - MultiCare Health System, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A SAD Cohort 1, 0.3 mg/kg ANK-700: All enrolled patients will receive one dose of 0.3 mg/kg ANK-700
  ANK-700: Intravenous (IV) infusion
- Part A SAD Cohort 2, 1.0 mg/kg ANK-700: All enrolled patients will receive one dose of 1.0 mg/kg ANK-700
  ANK-700: Intravenous (IV) infusion
- Part A SAD Cohort 3, 3.0 mg/kg ANK-700: All enrolled patients will receive one dose of 3.0 mg/kg ANK-700
  ANK-700: Intravenous (IV) infusion
- Part B MAD Cohort 4, 0.3 mg/kg ANK-700: All enrolled patients will receive three doses of 0.3 mg/kg ANK-700
  ANK-700: Intravenous (IV) infusion
- Part B MAD Cohort 5, 1.0 mg/kg ANK-700: All enrolled patients will receive three doses of 1.0 mg/kg ANK-700
  ANK-700: Intravenous (IV) infusion
- Part B MAD Cohort Placebo: All enrolled patients will receive three doses of Placebo
  Placebo: Intravenous (IV) infusion
Period: Overall Study
Arm/Group | Part A SAD Cohort 1, 0.3 mg/kg ANK-700 | Part A SAD Cohort 2, 1.0 mg/kg ANK-700 | Part A SAD Cohort 3, 3.0 mg/kg ANK-700 | Part B MAD Cohort 4, 0.3 mg/kg ANK-700 | Part B MAD Cohort 5, 1.0 mg/kg ANK-700 | Part B MAD Cohort Placebo
Started | 3 | 3 | 3 | 9 | 8 | 8
Completed | 3 | 3 | 3 | 9 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A SAD Cohort 2, 1.0 mg/kg ANK-700 | Part A SAD Cohort 1, 0.3 mg/kg ANK-700 | Part A SAD Cohort 3, 3.0 mg/kg ANK-700 | Part B MAD Cohort 4, 0.3 mg/kg ANK-700 | Part B MAD Cohort 5, 1.0 mg/kg ANK-700 | Part B MAD Cohort Placebo | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9 | 8 | 8 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 9 | 8 | 8 | 34
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (7.00) | 50.3 (6.43) | 48.7 (9.87) | 49.1 (8.43) | 50.9 (7.49) | 44 (9.59) | 48.2 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 7 | 7 | 6 | 24
  Male | 2 | 3 | 0 | 2 | 1 | 2 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 1 | 0 | 3
  White | 1 | 3 | 3 | 7 | 7 | 8 | 29
  Mixed | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing | 1 | 0 | 0 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 9 | 8 | 8 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Incidence and severity of treatment-emergent adverse events (TEAEs) as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 or higher
Time Frame: Up to 1 year
Population: All patients who received any amount of study drug with treatment group based on the dose level received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A SAD Cohort 1, 0.3 mg/kg ANK-700 | Part A SAD Cohort 2, 1.0 mg/kg ANK-700 | Part A SAD Cohort 3, 3.0 mg/kg ANK-700 | Part B MAD Cohort 4, 0.3 mg/kg ANK-700 | Part B MAD Cohort 5, 1.0 mg/kg ANK-700 | Part B MAD Cohort Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 9 | 8 | 8
Participants
  TEAE | 2 | 1 | 3 | 9 | 6 | 6
  Grade 3 or higher TEAE | 1 | 0 | 0 | 3 | 1 | 1
  SAE | 1 | 0 | 0 | 1 | 1 | 0
  no TEAE | 1 | 2 | 0 | 0 | 2 | 2

2. Secondary Outcome: CMAX
Description: Geometric mean of maximum plasma concentration (Cmax)
Time Frame: Days 1 and 7: One PK sample was taken pre-dose (≥at least 5 min prior to infusion), with all subsequent PK samples taken after end of infusion at the following time points: 0 min, 7min, 15min, 30min, 1h, 2h, 3h, 4h, 6h, 8h
Population: PK Analysis Set (PKAS) included all enrolled patients who received ≥ 1 complete dose of study drug and had ≥ 1 pre-dose and 1 post-dose measurement.
Measure: Geometric Mean (Full Range); unit: ng/mL
Groups:
- Part B MAD Cohort 4, 0.3 mg/kg ANK-700ANK-700: All enrolled patients will receive three doses of 0.3 mg/kg ANK-700
  ANK-700: Intravenous (IV) infusion
Arm/Group | Part A SAD Cohort 1, 0.3 mg/kg ANK-700 | Part A SAD Cohort 2, 1.0 mg/kg ANK-700 | Part A SAD Cohort 3, 3.0 mg/kg ANK-700 | Part B MAD Cohort 4, 0.3 mg/kg ANK-700ANK-700 | Part B MAD Cohort 5, 1.0 mg/kg ANK-700
Number analyzed (Participants) | 2 | 3 | 2 | 8 | 8
ng/mL
  Day 1 | NA [1308 to 1349] — not applicable; insufficient number of samples to calculate | 7120.7 [3380 to 12096] | NA [20462 to 33374] — not applicable; insufficient number of samples to calculate | 800.28 [105 to 1448] | 3816 [1830 to 9760]
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 8 | 5
  Day 7 |  |  |  | 540.99 [42.6 to 1650] | 1942.2 [197 to 9570]

3. Secondary Outcome: AUC Last
Description: Area under the plasma concentration-time curve from time 0 to the last measurable time point (AUC last)
Time Frame: Days 1 and 7: One PK sample was taken pre-dose (≥at least 5 min prior to infusion), with all subsequent PK samples taken after the end-of-infusion at the following time points: 0 min, 7 min, 15min, 30 min, 1h, 2h, 3h, 4h, 6h, 8h
Population: as for outcome 2
Measure: Geometric Mean (Full Range); unit: h*ng/mL
Arm/Group | Part A SAD Cohort 1, 0.3 mg/kg ANK-700 | Part A SAD Cohort 2, 1.0 mg/kg ANK-700 | Part A SAD Cohort 3, 3.0 mg/kg ANK-700 | Part B MAD Cohort 4, 0.3 mg/kg ANK-700ANK-700 | Part B MAD Cohort 5, 1.0 mg/kg ANK-700
Number analyzed (Participants) | 2 | 3 | 2 | 8 | 8
h*ng/mL
  Day 1 | NA [431 to 488] — not applicable; insufficient number of samples to calculate | 3620 [1530 to 6270] | NA [13600 to 19800] — not applicable; insufficient number of samples to calculate | 309 [45.1 to 551] | 1620 [529 to 4480]
  Day 7: number analyzed (Participants) | 0 | 0 | 0 | 8 | 5
  Day 7 |  |  |  | 217 [16.2 to 661] | 887 [149 to 4700]

ADVERSE EVENTS:
Time Frame: Up to 393 days (1 year + 28 days screening period)
Groups:
- MAD Cohort 4, 0.3 mg/kg ANK-700: All enrolled patients will receive three doses of 0.3 mg/kg ANK-700
  ANK-700: Intravenous (IV) infusion
- MAD Cohort 5, 1.0 mg/kg ANK-700: All enrolled patients will receive three doses of 1.0 mg/kg ANK-700
  ANK-700: Intravenous (IV) infusion
- MAD Cohort Placebo: All enrolled patients will receive three doses of Placebo
  Placebo: Intravenous (IV) infusion
Arm/Group | ANK-700 SAD Cohort 1, 0.3 mg/kg ANK-700 | ANK-700 SAD Cohort 2, 1.0 mg/kg ANK-700 | ANK-700 SAD Cohort 3, 3.0 mg/kg ANK-700 | MAD Cohort 4, 0.3 mg/kg ANK-700 | MAD Cohort 5, 1.0 mg/kg ANK-700 | MAD Cohort Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/9 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 1/9 | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 3/3 | 9/9 | 6/8 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANK-700 SAD Cohort 1, 0.3 mg/kg ANK-700 (N=3) | ANK-700 SAD Cohort 2, 1.0 mg/kg ANK-700 (N=3) | ANK-700 SAD Cohort 3, 3.0 mg/kg ANK-700 (N=3) | MAD Cohort 4, 0.3 mg/kg ANK-700 (N=9) | MAD Cohort 5, 1.0 mg/kg ANK-700 (N=8) | MAD Cohort Placebo (N=8)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANK-700 SAD Cohort 1, 0.3 mg/kg ANK-700 (N=3) | ANK-700 SAD Cohort 2, 1.0 mg/kg ANK-700 (N=3) | ANK-700 SAD Cohort 3, 3.0 mg/kg ANK-700 (N=3) | MAD Cohort 4, 0.3 mg/kg ANK-700 (N=9) | MAD Cohort 5, 1.0 mg/kg ANK-700 (N=8) | MAD Cohort Placebo (N=8)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (7) | 1 (2) | 1 (2)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple Sclerosis relapse (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Multiple Sclerosis pseudo relapse (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gait spastic (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site discolouration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac checst pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phsophatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza A virus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte percentage decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Facial myokymia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depersonalisation/derealization disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Middle insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT04602390/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT04602390/SAP_001.pdf